CLINICAL TRIAL: NCT04788485
Title: Evaluation of Smectite Effect As A Food Thickener On Gastroesophageal Reflux Disease In Neonates Using Combined Esophageal Multichannel Intraluminal Impedance
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Hend Fayez Ahmed, specialist, Ain Shams Maternity Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: PH-MII in neonates
Record Dates: First submitted 2021-03-05; First posted 2021-03-09 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Gastroesophageal Reflux in Neonates
MeSH Terms: interventions — Smectite; smecta

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Neonates before adding smectite (Active Comparator): neonates will receive diosmectite for treating of gastroesophageal reflux in neonates after MII-ph
  Interventions: Drug: Diosmectite
- neonates after adding smectite (Active Comparator): neonates after they received diosmectite for treating of gastroesophageal reflux in neonates after MII-ph
  Interventions: Drug: Diosmectite

INTERVENTIONS:
Drug: Diosmectite — use of diosmectite as a food thickener in neonates in with gastroesophageal reflux in noenates
  Other Names: Smecta

SUMMARY:
study of diagnosis of GERD in neonates by MII-PH with trial of smectite for treatment

DETAILED DESCRIPTION:
This is a prospective clinical trial conducted on 20 preterm neonates < 37 weeks of gestation, admitted in NICU, maternity hospital, Ain Shams University. They were assessed for gastroesophageal reflux disease and investigated using ph-MII for detection of reflux episodes and they were given Smecta 3gm/day for 7 days at least as a food thickener and then ph-MII repeated to assess the response

ELIGIBILITY:
Inclusion Criteria:

* • Newborns free of any congenital anomalies or inborn errors of metabolism

  * Infants had signs of reflux like:

    1. Typical or atypical crying and/or irritability
    2. Apparent life-threatening event
    3. Poor appetite; weight loss or poor growth (failure to thrive)
    4. Vomiting
    5. Bronchopulmonary dysplasia
    6. Wheezing, stridor
    7. Recurrent pneumonitis
    8. Sandifer syndrome (ie, posturing with opisthotonus or torticollis)

Exclusion Criteria:

* • Newborns with GIT anomalies as trans-esophageal fistula, hiatus hernia and other GIT anomalies causing reflux.

  * Patients with Hirshsprung disease or delayed passage of meconium.
  * History of NEC in the baby.

Ages: 0 Days to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2021-02-25 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Effect of smectite as food thickener for treatment of gastroesophgeal reflux in neonates | within 7 days
  efficacy of Smectite as a food thickener in treating GERD in neonates using Multichannel intraluminal impedance-pH monitoring.

SECONDARY OUTCOMES:
Reliability of signs for diagnosis of gastroesophageal reflux in neonates using MII-pH | within 24 hours
  determine the reliability of signs such as cardio-respiratory events, apneas and dystonic neck posturing (Sandifer syndrome) in the diagnosis of GERD using Multichannel intraluminal impedance-pH monitoring.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University-Faculty of Medicine, Cairo, Egypt